CLINICAL TRIAL: NCT07047820
Title: Prospective, Observational Survey Study Assessing Effectiveness of Zuranolone in Improving PPD Symptoms in the Real-world Setting
Brief Title: A Study to Learn More About How Zuranolone Affects Postpartum Depression Symptoms in Participants Who Took it Within 1 Year After The End of Their Pregnancy
Status: Recruiting | Type: Observational
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: US-ZRN-12349
Record Dates: First submitted 2025-06-25; First posted 2025-07-02 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Depression, Postpartum
MeSH Terms: conditions — Depression, Postpartum | interventions — zuranolone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Zuranolone: Participants who are prescribed zuranolone for PPD and are filling zuranolone through a consumer value store (CVS) specialty pharmacy will be contacted through email or the call center for enrollment in the study.
  Interventions: Drug: Zuranolone

INTERVENTIONS:
Drug: Zuranolone — Administered as specified in the treatment arm
  Other Names: Zurzuvae; BIIB125

SUMMARY:
In this study, researchers will learn more about how zuranolone affects the symptoms of postpartum depression, also known as PPD. Zuranolone is a drug that healthcare professionals can prescribe for adults with PPD. After giving birth, adults with PPD can suffer from symptoms such as tiredness, sadness, and a loss of interest in their daily activities.

This study is known as an observational study, which means it collects health information about study participants after a healthcare professional has already prescribed treatment. Participants for this study will be found in the United States using a database from CVS Specialty Pharmacy. This will include anyone who was prescribed zuranolone between June 2025 and May 2026 and who filled the prescription within 1 year after the end of their pregnancy.

The main goal of this study is to learn more about how zuranolone affects the participants' PPD symptoms. This will be measured using a questionnaire completed by participants called the Edinburgh Postnatal Depression Scale, also known as the EPDS. A higher score on the EPDS may indicate more severe PPD symptoms.

The main question researchers want to answer in this study is:

- Do PPD symptoms change after treatment with zuranolone based on EPDS scores measured at Day 15?

Researchers will also learn more about:

* Changes in participants' EPDS scores from before treatment to Day 45, which is 30 days after treatment ends.
* How many participants breastfeed their babies while taking zuranolone
* How many participants do not start new medicine after finishing their zuranolone treatment
* How many participants take new medicines after finishing zuranolone
* How many participants already tried other medicines for their depression symptoms before joining this study
* How many participants take other medicines in general while taking zuranolone

This study will be done as follows:

People who fill their zuranolone prescription through CVS Specialty Pharmacy will be contacted by email or phone to ask them about their interest in participating in the study.

Those who agree to take part will answer written questions about their symptoms using the EPDS tool. They will also answer other survey questions about their background, environment, and general health information. Participants must take their first dose of zuranolone within 7 days of joining the study.

Participants will then be asked to answer questions using the EPDS tools, 15 days and 45 days after taking the first dose of zuranolone.

DETAILED DESCRIPTION:
The primary objective of this study is to assess the effectiveness of zuranolone in reducing postpartum depression (PPD) symptoms via the Edinburgh Postnatal Depression Scale (EPDS) at Day 15. The secondary objectives are to assess the effectiveness of zuranolone in reducing PPD symptoms via the EPDS at Day 15 and Day 45 in a subgroup of participants with moderate PPD at baseline, in reducing PPD symptoms via the EPDS at Day 45, to assess breastfeeding status during treatment with zuranolone at Day 45 and to characterize treatment usage across the 45-day period via self-reported survey questions.

ELIGIBILITY:
Key Inclusion Criteria:

* Adults who were prescribed and had one successful fill for zuranolone within 12 months following end of pregnancy for the treatment of PPD from June 2025 to May 2026 through CVS Specialty Pharmacy.
* Currently reside in the United States.
* Able to complete the questionnaires independently.

Key Exclusion Criteria:

* Prior fill of zuranolone or brexanolone in last 12 months.
* Participants with 2 or more doses of zuranolone at the time of screening.
* Current or history of bipolar disorder.
* Failure to complete baseline surveys prior to 2nd dose of zuranolone.
* Pregnancy that ended more than 12 months ago.

Other protocol-defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Participants prescribed zuranolone who consent to participate in this study and meet all of the inclusion criteria, none of the exclusion criteria, and complete baseline (Day 0) will be considered enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2026-08-24 (Estimated); Study Completion 2026-08-24 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Edinburgh Postnatal Depression Scale (EPDS) at Day 15 | Baseline (Day 0), Day 15
  EPDS is a 10-item self-report questionnaire used for the assessment of PPD symptoms. Each item is scored from 0-3, with a total score range of 0-30. Higher scores indicate more severe depressive symptoms.

SECONDARY OUTCOMES:
Change From Baseline in EPDS at Day 45 | Baseline (Day 0), Day 45
  EPDS is a 10-item self-report questionnaire used for the assessment of PPD symptoms. Each item is scored from 0-3, with a total score range of 0-30. Higher scores indicate more severe depressive symptoms.
Change From Baseline in EPDS in Participants With Moderate Postpartum Depression (PPD) Severity at Days 15 and 45 | Baseline (Day 0), Days 15 and 45
  EPDS is a 10-item self-report questionnaire used for the assessment of PPD symptoms. Each item is scored from 0-3, with a total score range of 0-30. Higher scores indicate more severe depressive symptoms.
Number of Participants That Self-Report no New Initiation of Medication After Completion of Zuranolone | Day 45
Number of Participants With Moderate PPD Severity That Self-Report no New Initiation of Medication After Completion of Zuranolone | Day 45
Number of Participants That Self-Report Feeding Their Baby Breastmilk as Usual While Taking Zuranolone | Day 45
Number of Participants That Self-Report History of Medication Use for Depression | Day 0
Number of Participants With Moderate PPD Severity That Self-Report History of Medication Use for Depression | Day 0
Number of Participants That Self-Report Prior Lines of Treatment for Their Current PPD Episode | Day 0
Number of Participants With Moderate PPD Severity That Self-Report Prior Lines of Treatment for Their Current PPD Episode | Day 0
Number of Participants That Self-Report Concomitant Medication Use With Zuranolone for the Treatment of PPD | Day 0
Number of Participants With Moderate PPD Severity That Self-Report Concomitant Medication Use With Zuranolone for the Treatment of PPD | Day 0

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- CVS Health, Woonsocket, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on htps://www.biogentrialtransparency.com/
URL: https://vivli.org/